CLINICAL TRIAL: NCT04264598
Title: A Phase I Study to Evaluate the Safety and Immunogenicity of a Sabin Inactivated Poliovirus Vaccine (Vero Cell)
Brief Title: Safety and Immunogenicity of a Sabin Inactivated Poliovirus Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Collaborators: Beijing Minhai Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2017L00935
Record Dates: First submitted 2020-02-09; First posted 2020-02-11 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Polio
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Experimental Adult Group - Medium dosage (Experimental): One intramuscular injection of the investigational vaccine (0.5 ml); Intervention: one-dose regimen of medium dosage investigational sIPV Intervention: Biological: one-dose regimen of medium dosage investigational sIPV
  Interventions: Biological: sIPV
- Experimental Children Group - Medium dosage (Experimental): One intramuscular injection of the investigational vaccine (0.5 ml); Intervention: one-dose regimen of medium dosage investigational sIPV Intervention: Biological: one-dose regimen of medium dosage investigational sIPV
  Interventions: Biological: sIPV
- Experimental Infant Group - Medium dosage (Experimental): Three intramuscular injections of the investigational vaccine (0.5 ml) on Day 0, Day 30 and Day 60 respectively; Intervention: Three-dose regimen of medium dosage investigational sIPV Intervention: Biological: Three-dose regimen of medium dosage investigational sIPV
  Interventions: Biological: sIPV
- Control Infant Group - commercialized sIPV (Active Comparator): Three intramuscular injections of the investigational vaccine (0.5 ml) on Day 0, Day 30 and Day 60 respectively; Intervention: Three-dose regimen of commercialized sIPV Intervention: Biological: Three-dose regimen of commercialized sIPV
  Interventions: Biological: Commercialized sIPV
- Control Infant Group - commercialized IPV (Active Comparator): Three intramuscular injections of the investigational vaccine (0.5 ml) on Day 0, Day 30 and Day 60 respectively; Intervention: Three-dose regimen of commercialized IPV Intervention: Biological: Three-dose regimen of commercialized IPV
  Interventions: Biological: Commercialized IPV

INTERVENTIONS:
Biological: sIPV — The Medium dosage sIPV was developed by Minhai Biotech Co., LTD. The antigen contents of type I, type II and type III polioviruses in the medium dosage sIPV were 15 DU, 45 DU and 45 DU. The vaccine was in liquid form, 0.5 ml per dose.
  Arms: Experimental Adult Group - Medium dosage; Experimental Children Group - Medium dosage; Experimental Infant Group - Medium dosage
Biological: Commercialized sIPV — The commercialized sIPV was manufactured by Institute of Medical Biology Chinese Academy of Medical Sciences.The antigen contents of type I, type II and type III polioviruses in the commercialized sIPV were 30 DU, 32 DU and 45 DU. The vaccine was in liquid form, 0.5 ml per dose.
  Arms: Control Infant Group - commercialized sIPV
Biological: Commercialized IPV — The commercialized Salk IPV was manufactured by Sanofi Pasteur S.A.The antigen contents of type I, type II and type III polioviruses in the commercialized IPV were 40 DU, 8 DU and 32 DU. The vaccine was in liquid form, 0.5 ml per dose.
  Arms: Control Infant Group - commercialized IPV

SUMMARY:
The purpose of this phase I study is to evaluate the safety of a Sabin Inactivated Poliovirus Vaccine (sIPV) in adults and children, and the safety and immunogenicity of it in infants. 20 adults aged 18~45 years and 20 children aged 4 years were only administered one dose of sIPV with medium D antigen content. 60 infants aged 2 months (60~90 days) were randomized to receive three doses of sIPV with medium D antigen content, conventional IPV (cIPV, manufactured by Sanofi Pasteur) or sIPV (manufactured by the Institute of Medical Biology, the Chinese Academy of Medical Biology), respectively, on the month 0, 1, 2 schedule. Serum samples were collected before the 1st dose and 30 days after the 3rd dose vaccination to assess the immunogenicity in infants. Adverse events occurring within 30 days after each dose were collected to assess the safety.

DETAILED DESCRIPTION:
The purpose of this phase I study is to evaluate the safety of a Sabin Inactivated Poliovirus Vaccine (sIPV) in adults and children, and the safety and immunogenicity of it in infants. 20 adults aged 18~45 years and 20 children aged 4 years were only administered one dose of sIPV with medium D antigen content. 60 infants aged 2 months (60~90 days) were randomized to receive three doses of sIPV with medium D antigen content, conventional IPV (cIPV, manufactured by Sanofi Pasteur) or sIPV (manufactured by the Institute of Medical Biology, the Chinese Academy of Medical Biology), respectively, on the month 0, 1, 2 schedule. Serum samples were collected before the 1st dose and 30 days after the 3rd dose vaccination to assess the immunogenicity in infants. Adverse events occurring within 30 days after each dose were collected to assess the safety.

The antigen contents of type I, type II and type III polioviruses in the investigational and control vaccines were as follows: medium-dose Sabin IPV (15 DU, 45 DU and 45 DU), control Sabin IPV (30 DU, 32 DU and 45 DU), control Salk IPV (40 DU, 8 DU and 32 DU). All vaccines were in liquid form, 0.5 ml per dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer aged 18~45 years with/without prior vaccination of poliovirus and without any contraindication for vaccination;
* Healthy volunteer aged 4 years with/without prior vaccination of poliovirus but without booster vaccination and any contraindication for vaccination;
* Healthy volunteer aged 2 months (60~90 days) without prior vaccination of poliovirus and any contraindication for vaccination;
* Guardians of the participants should be capable of understanding the written consent form, and such form should be signed prior to enrolment;
* Complying with the requirement of the study protocol;
* Axillary temperature ≤ 37.0 °C;

Exclusion Criteria:

* Women aged 18~45 years with positive urine pregnancy test, pregnant or lactating women, or women with pregnancy plans within 3 months;
* Preterm or low birth weight infants;
* Congenital malformation, developmental disorders, genetic defects, or severe malnutrition;
* History of polio;
* Severe nervous system disease (epilepsy, seizures or convulsions) or mental illness;
* History of allergy to any vaccine, or any ingredient of the vaccine, or serious adverse reaction(s) to vaccination, such as urticaria, dyspnea, angioneurotic edema, abdominal pain, etc;
* Autoimmune disease or immunodeficiency/immunosuppressive;
* Bleeding disorder diagnosed by a doctor (e.g., coagulation factor deficiency, coagulation disorder, or platelet disorder), or significant bruising or coagulopathy;
* Serious chronic diseases, respiratory diseases, cardiovascular diseases, liver or kidney diseases or skin diseases;
* Mother of the participant has HIV infection;
* Acute illness or acute exacerbation of chronic disease within the past 7 days;
* Had a high fever within the past 3 days (axillary temperature ≥ 38.0°C);
* Receipt of any subunit or inactivated vaccine within the past 7 day;
* Receipt of any live attenuated vaccine within the past 14 days;
* Receipt of any blood product within the past 3 months;
* Any other factor that, in the judgment of the investigator, suggesting the volunteer is unsuitable for this study;

Ages: 60 Days to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2017-12-19 (Actual); Study Completion 2018-12-28 (Actual)

PRIMARY OUTCOMES:
The seroconversion rates (SCRs) of each group 30 days after three-dose regimen | 28~42 days
  Subjects whose pre-immune antibody level < 1:8 and post-immune antibody level ≥ 1:8, or those whose pre-immune antibody level ≥ 1:8 and the increase of post-immune antibody level ≥ 4 folds are considered seroconverted.

SECONDARY OUTCOMES:
The geometric mean titer (GMT) of each group 30 days after three-dose regimen | 28~42 days
  GMT of each group 28~42 days after three-dose regimen.
The geometric mean fold increase (GMI) of each group 30 days after three-dose regimen | 28~42 days
The number of participants who have adverse reactions divided by the total number of participants | 30 days
The number of participants who have adverse events (AEs) divided by the total number of participants. | 30 day
  occurred within 30 days after each injection

CONTACTS AND LOCATIONS:
Overall Officials: Fengcai Zhu, Master, Principal Investigator — Jiangsu Provincial Center for Disease Control and Prevention
Locations (1):
- Jiangsu Provincial Center for Diseases Control and Prevention, Nanjing, China

REFERENCES:
- [Derived] Jia S, Tang R, Li G, Hu Y, Liang Q. The effect of maternal poliovirus antibodies on the immune responses of infants to poliovirus vaccines. BMC Infect Dis. 2020 Aug 31;20(1):641. doi: 10.1186/s12879-020-05348-1. PMID 32867698